CLINICAL TRIAL: NCT04361487
Title: Circumferential Compression STITCH Repairs of Complex and Horizontal Cleavage Meniscal Tears
Acronym: NOVOSTITCH PRO
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NOVOSTITCH.2019.09
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-11

CONDITIONS: Meniscus Tear; Retention; Meniscus
Keywords: NOVOSTITCH; meniscal; meniscus; repair; knee; horizontal cleavage; complex tear; arthroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Horizontal Cleavage Meniscal Tear: Participants with horizontal cleavage meniscal tears
  Interventions: Device: NOVOSTITCH PRO Meniscal Repair System
- Complex Meniscal Tear: Participants with complex meniscal tears
  Interventions: Device: NOVOSTITCH PRO Meniscal Repair System

INTERVENTIONS:
Device: NOVOSTITCH PRO Meniscal Repair System — Standard of care surgery with in which the meniscus is repaired using NOVOSTITCH PRO

SUMMARY:
The purpose of this study is to understand the benefits and safety of the NOVOSTITCH PRO Meniscal Repair (NOVOSTITCH PRO) system. The meniscus is a tissue in the knee joint. The NOVOSTITCH PRO is used during surgery to fix meniscus tears in the knee. It is unknown whether fixing a meniscus tear is better than the approach of removing the tear. Data will be collected on participants prior to surgery, at surgery, and for 2 years after surgery.

DETAILED DESCRIPTION:
The purpose of this study is to understand the benefits and safety of the NOVOSTITCH PRO Meniscal Repair (NOVOSTITCH PRO) system. The meniscus is a tissue in the knee joint. The NOVOSTITCH PRO is used during surgery to fix meniscus tears in the knee. It is unknown whether fixing a meniscus tear is better than the approach of removing the tear. Data will be collected on participants prior to surgery, at surgery, and for 2 years after surgery.

There are different types of tears in the meniscus. This study includes 2 of the tear types: horizontal cleavage and complex meniscal tears.

Participants will be consented and enrolled in the study prior to knee surgery. Participants will complete surveys before surgery and data obtained from the medical record. In addition, standard of care x-rays and MRIs of the knee will be sent to the study. Participants will have their standard of care surgery to repair the knee using NOVOSTITCH PRO. Images and videos inside the knee during surgery may be sent to the study.

Participants will be followed 2 years after surgery. There are a total of 5 follow-up visits: 2 weeks, 3 months, 6 months, 1 year, and 2 years after surgery. Data will be obtained from medical records, surveys, MRIs, and radiographs. Up to 30 participants will have an optional needle endoscopy at the 6-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible for the study if they meet all of the following criteria at the Baseline Screening:

  1. Able and willing to give informed consent by voluntarily providing written informed consent in accordance with governing Institutional Review Board;
  2. 18 to 70 years of age, inclusive at the time of screening;
  3. History indicative of meniscal pathology (e.g., pain, mechanical symptoms described as locking, clicking or giving way);
  4. Physical exam consistent with meniscus tear (e.g., locked joint, joint line tenderness and/or pain on meniscal compression);
  5. If prior ligament reconstruction, the study knee is clinically stable;
  6. Meniscal repair to be performed arthroscopically;
  7. Preoperative MRI evidence consistent with a horizontal cleavage or complex meniscus tear in the symptomatic compartment;
  8. Willing and able to comply with all study procedures and visit requirements, including MRIs, X-rays, and Case Report Forms (CRFs) completed by the subject.
* Consented subjects may be included in the study only if, upon arthroscopic inspection during the procedure, their meniscal study lesion meets all of the following criteria:

  1. Meniscal tear amenable to repair with NOVOSTITCH PRO with or without the use of adjunct devices per the exclusion criteria;
  2. Tear pattern is one of the following:

     1. Horizontal cleavage tear (HCT), or
     2. Complex multi-planar tear (combination of at least two of the following tears: horizontal, oblique, radial, vertical).

Exclusion Criteria:

* Subjects will be excluded from the study if they meet any of following criteria at the Baseline Screening:

  1. Arthritis in the study knee (Kellgren-Lawrence Grade 3 or higher);
  2. Body Mass Index (BMI) ≥40 kg/m2;
  3. Previous surgical meniscal repair or meniscectomy of the study meniscus;
  4. Unstable knee;
  5. Clinically significant malalignment of the study knee, and/or requiring osteotomy, and/or correction;
  6. History of constitutional/systemic inflammatory/arthritic problem or pain condition, history of knee infection, vascular condition of legs, benign neoplasms of knee, hepatitis, and/or HIV;
  7. Currently on any immunosuppressive therapy;
  8. Expected to undergo any other surgical treatment of either knee;
  9. Previously enrolled in the study (no bilateral knee surgeries);
  10. Surgical procedures other than those listed in the Indications for Use;
  11. Patient conditions including insufficient quantity or quality of tissue;
  12. Insufficient blood supply or previous infections which may hinder the healing process;
  13. Foreign body sensitivity. If material sensitivity is suspected, testing should be completed prior to suture implantation;
  14. Conditions which may limit the patient's ability or willingness to follow postoperative care instructions;
  15. Any concomitant painful or disabling disease, condition or post-procedure status of either lower extremity that would interfere with evaluation or rehabilitation of the study knee;
  16. Pregnant or planning to become pregnant in the next 2 years;
  17. Subject does not understand a language in which the PROs and EQ-5D-5L are available.
* Subjects will be excluded from the study if their study meniscus lesion meets any of the following criteria at arthroscopy:

  1. Ramp tears;
  2. Root or other tear type requiring tibial fixation;
  3. Tears requiring repair of both meniscus in the study knee;
  4. Intact or partially intact meniscus tear that, in the opinion of the Investigator, does not require repair;
  5. Poor meniscal tissue quality such that it will not hold a suture;
  6. For HCTs:

     1. Use of any capsular fixation device; OR
     2. Any portion of the meniscal tear is repaired using a device to place stitches other than NOVOSTITCH PRO, Meniscus Mender II, or Meniscal Stitcher, or FIRSTPASS MINI marketed by Smith + Nephew Inc.;
  7. For complex tears:

     a. Any portion of the meniscal tear is repaired using a device to place stitches other than NOVOSTITCH PRO, Meniscus Mender II, Meniscal Stitcher, FIRSTPASS MINI, FAST-FIX 360, or ULTRA FAST-FIX marketed by Smith + Nephew Inc.;
  8. Clinically significant (zone 1 and/or zone 2) tear in the contralateral compartment to the study meniscus;
  9. Performance of a significant concomitant procedure (e.g. ACL reconstruction or repair, cartilage repair or restoration) intended as a therapeutic intervention on the study knee;
  10. Presence of infection;
  11. Articular cartilage damage in the study knee, defined as Modified Outerbridge Grade III or higher.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited at the sports medicine/orthopedic clinic.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of reoperation due to meniscal repair failure at 12 months after surgery | 12 months

SECONDARY OUTCOMES:
Rate of reoperation due to meniscal repair failure at 6 months after surgery | 6 months
Rate of reoperation due to meniscal repair failure at 24 months after surgery | 24 months
Structural integrity of meniscus assessed by MRI | 12 and 24 months
Tibiofemoral joint space narrowing assessed by x-ray | 12 months
Healing status assessed by in-office needle endoscopy | 6 months
Patient Reported Outcome (PRO): International Knee Documentation Committee (IKDC) Subjective ScoreOutcomes scores | 6, 12, and 24 months
  The International Knee Documentation Committee (IKDC) Subjective score was developed to detect improvement or deterioration in symptoms, function, and sports activities due to knee impairment, including patients with meniscal injuries.
  There are three domains: 1) symptoms, including pain, stiffness, swelling, locking/catching, and giving way (7 items), 2) sports and daily activities (10 items), and 3) current knee function and knee function prior to knee injury (1 item, not included in the score). Responses vary for each item. The possible score ranges from 0-100, where 100 = no limitation with daily or sporting activities and the absence of symptoms.
Patient Reported Outcome (PRO): Knee Injury and Osteoarthritis Outcome Score (KOOS) Outcomes scores | 6, 12, and 24 months
  There are five patient-relevant subscales of the KOOS, and each are scored separately:
  Pain (9 items), Symptoms (7 items), ADL function (17 items), Sport and Recreation Function (5 items), and Quality of Life (4 items).
  A Likert scale is used and all items have five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the 5 scores is calculated as the sum of the items included and then each score is transformed to a 0-100 scale, with 0 representing extreme knee problems and 100 representing no knee problems as common in orthopedic assessment scales and generic measures. An aggregate score is not calculated so that each of the 5 dimensions can be assess separately.
Patient Reported Outcome (PRO):LysholmOutcomes scores | 6, 12, and 24 months
  This tool measures the domains of symptoms and complaints and functioning of daily activities. The scale consists of 8 item and is scaled from 0 to 100, with a higher score indicating fewer symptoms and higher level of functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Karlie Morgan, BS CCRP, Study Chair — Smith & Nephew, Inc.
Locations (6):
- United States (6):
  - CAO Research Foundation, Washington D.C., District of Columbia
  - Hawai'i Pacific Health / Straub Medical Center, Honolulu, Hawaii
  - Rush University Medical Center / Midwest Orthopaedics at Rush, Chicago, Illinois
  - University of Kansas Medical Center, Overland Park, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - Ohio State University/Jameson Crane Sports Medicine Institute, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No